CLINICAL TRIAL: NCT04296344
Title: Group Acupuncture Therapy With Modified Yoga for Chronic Neck, Low Back and OA Pain in Safety Net Setting for an Underserved Population (GAPYOGA)
Brief Title: Group Acupuncture Therapy With Modified Yoga
Acronym: GAPYOGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: The Institute for Family Health (Other); Albert Einstein College of Medicine (Other); Maryland University of Integrative Health (Other)
Responsible Party: Principal Investigator, Raymond Teets, Assistant Professor, Family Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 18-1240; 02855405 (Other Grant/Funding Number: Blavatnik Family Foundation)
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Chronic Neck Pain; Chronic Low Back Pain; Osteoarthritis Pain
Keywords: Acupuncture therapy; Yoga therapy; Integrative medicine; Chronic pain; Underserved; Safety net setting
MeSH Terms: conditions — Chronic Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Participants with chronic pain to receive acupuncture therapy treatments and yoga therapy sessions.
  Interventions: Other: Acupuncture Therapy Treatments; Other: Yoga Therapy Sessions

INTERVENTIONS:
Other: Acupuncture Therapy Treatments — 10 consecutive weekly group acupuncture therapy treatments
Other: Yoga Therapy Sessions — 8 consecutive yoga therapy sessions that occur immediately following in a room adjacent to acupuncture therapy.

SUMMARY:
Chronic pain is prevalent in the U.S., with impact on physical and psychological functioning as well as lost work productivity. Minority and lower socioeconomic populations have increased prevalence of chronic pain with less access to pain care and poorer outcomes. Acupuncture therapy is effective in treating chronic pain conditions including chronic low back pain (cLBP), neck pain, shoulder pain and knee pain from osteoarthritis (OA). Acupuncture therapy, including group acupuncture, is feasible and effective, and specifically so for underserved and diverse populations at risk for health outcome disparities. Acupuncture therapy also encourages patient engagement and activation. As chronic pain improves there is a natural progression to want and need to increase activity and movement recovery. Diverse movement approaches are important both for improving range of motion, maintaining gains, strengthening and promoting patient engagement and activation. Yoga therapy is an active therapy with proven benefit in musculoskeletal pain disorders and pain associated disability. The aim of this pilot feasibility trial is to test the bundling of these two care options for chronic pain, to inform both the design for a larger randomized pragmatic effectiveness trial as well as implementation strategies across underserved settings.

DETAILED DESCRIPTION:
The goal of this project is to assess the feasibility of a low-cost, integrative intervention for chronic pain that can be replicated and implemented in underserved medical settings across the U.S. Over the course of 18 months, the study team will recruit at least 150 outpatients with chronic pain from the Institute for Family Health (IFH) Family Medicine sites and Montefiore Medical Group sites, both Federally Qualified Health Centers (FQHCs). Treatment will consist of ten consecutive weekly group acupuncture therapy treatments. Yoga therapy treatments will start at week three and will consist of eight consecutive yoga therapy sessions that occur immediately following in a room adjacent to acupuncture therapy. Sessions are bundled to facilitate attendance that might be affected by two separate trips a week for participation. The primary outcome will be pain interference and pain intensity. Secondary outcomes will be pain free days, depression, functional status, patient activation, and pain medication utilization. These will be used during the pre-intervention phase, during which patients are receiving usual care only, and compared to the period after patients receive the combined acupuncture and yoga sessions. Data will be collected for 10 days before acupuncture and yoga therapy, and up to 24 weeks following the end of treatment.

The study will use a 'multiple settings across baseline' quasi-experimental design. This is a repeated measures design, and each study participant will have multiple pre- and post-measures. The multiple pre-measurement points allows the study team to document and monitor what may be variable patterns of pain pre-intervention. This design optimizes feasibility and acceptability to patients and participating health centers while still generating meaningful outcome data. Specifically, the study team has not proposed randomization within the practices, rather allowing sites to offer the intervention to all patients with target diagnoses who meet eligibility criteria. To collect pre-acupuncture assessments of pain, the study team will include a 10 day intake run-in period prior to the initial acupuncture session that ensures treatment within a time frame that is consistent with typical time to appointments for many consultations.

ELIGIBILITY:
Inclusion Criteria:

* Patients 21 years of age or older
* Chronic pain (three months or more in duration) due to a qualifying diagnosis of back pain, neck pain, and/or osteoarthritis.
* Eligible patients must be receiving primary care at a participating IFH or Montefiore Medical Group site
* Participants must understand and be able to provide consent in English or Spanish
* Reliable contact phone numbers must be available to facilitate scheduling,
* Availability for up to 10 weekly consecutive treatments and
* Availability for follow-up data collection at 24 weeks

Exclusion criteria:

* Receipt of acupuncture treatment or yoga instruction/therapy in the 6 months prior to recruitment
* Pregnancy
* Severe psychiatric problems as assessed by the study team (e.g., chronic interpersonal problems, cognitive impairment or active psychosis that is uncontrolled by medication that precludes the ability to provide informed consent or complete the survey instruments)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Change in Brief Pain Inventory: Short Form | Baseline and Week 24
  The BPI is a nine-item measure which that asks patients to indicate how their pain influences function: select aspects of their everyday life including mood, walking, sleep and their ability to work over the past 24 hours, as well as the level and intensity of pain. This measure will be adapted for use by phone, modifying a question which asks participants to refer to a diagram of the body. total score from 0 to 10, with higher score indicating worse outcomes.

SECONDARY OUTCOMES:
Change in Pain Free Days | Baseline and Week 24
  Self-report measure to report the number of pain free days in the previous 2 weeks. This measure will be used pre- and post-intervention.
Change in Center for Epidemiological Studies - Depression Scale (CES-D) | Baseline and Week 24
  This is a well-validated, 20-item measure of depressive symptoms. This will be used both at the initiation treatment interview and the end of the study. Full score from 0- 20, with higher score indicating more symptomology.
Change in Altarum Consumer Engagement (ACE) | Baseline and Week 24
  A 12-item measure that assesses three domains of health engagement: commitment, informed choice, and navigation. The measure covers areas not included in other surveys and it is a good predictor of current health status, lifestyle health behaviors, medication adherence, and how likely it is that people will use tools to support their decisions. This measure will be adapted to include 8 of the 12 items on the questionnaire. Full scale from 0-100, higher score indicates higher consumer engagement.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS 10) | Baseline and Week 24
  A series of person-centered measures that evaluate and monitor physical, mental, and social health in adults and children. 10-item patient-reported questionnaire. standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.
Change in PROMIS Satisfaction with Participation in Social Roles (PROMIS-SF) | Baseline and Week 24
  is a 14-item measure that is part of the PROMIS Social Function. The measure refers to social roles, such as work and family responsibilities, and more discretionary social activities, such as leisure activity and relationships with friends. standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.
Change in Patient Global Impression of Change (PGIC) | Week 10 and Week 24
  Patient Global Impression of Change (PGIC) is a single question 7-point categorical scale that captures a patient's experience of treatment at follow-up points, after all sessions are completed. Full score from 0-7, with higher score indicating more improvement.
Change in Medication Utilization | Baseline and Week 24
  Participants will be asked to report their use of pain medications over the prior one-week period.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Teets, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (3):
- United States (3):
  - The Institute For Family Health, New York, New York
  - Montefiore Family Health Center, The Bronx, New York
  - Williamsbridge Family Practice Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.Any purpose.Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at (Link to be provided).

REFERENCES:
- [Derived] Anderson BJ, Meissner P, Mah DM, Nielsen A, Moonaz S, McKee MD, Kligler B, Milanes M, Guerra H, Teets R. Barriers and Facilitators to Implementing Bundled Acupuncture and Yoga Therapy to Treat Chronic Pain in Community Healthcare Settings: A Feasibility Pilot. J Altern Complement Med. 2021 Jun;27(6):496-505. doi: 10.1089/acm.2020.0394. Epub 2021 Mar 15. PMID 33720749